CLINICAL TRIAL: NCT03555149
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Metastatic Colorectal Cancer (Morpheus-CRC)
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Metastatic Colorectal Cancer (Morpheus-CRC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor made the decision to terminate the study due to start up and recruitment issues caused by limited resource availability at the treating centers.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO39612; 2017-004566-99 (EudraCT Number)
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; atezolizumab; Bevacizumab; isatuximab; selicrelumab; RG7388

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Regorafenib (Control) (Active Comparator): Participants will receive treatment until unacceptable toxicity or disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
  Interventions: Drug: Regorafenib
- Atezolizumab + Imprime PGG + Bevacizumab (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Imprime PGG; Drug: Bevacizumab
- Atezolizumab + Isatuximab (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Isatuximab
- Atezolizumab + Selicrelumab + Bevacizumab (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Selicrelumab
- Atezolizumab + Idasanutlin (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Idasanutlin
- Atezolizumab + Regorafenib (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Regorafenib; Drug: Atezolizumab
- Atezolizumab + Regorafenib + AB928 (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Regorafenib; Drug: Atezolizumab; Drug: AB928
- Atezolizumab + LOAd703 (Experimental): Participants will receive treatment until unacceptable toxicity or loss of clinical benefit as confirmed by disease progression per RECIST V1.1 or lack of continued benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Genetic: LOAd703

INTERVENTIONS:
Drug: Regorafenib — Regorafenib will be administered orally on Days 1-21 of each 28-day cycle.
  Arms: Atezolizumab + Regorafenib; Atezolizumab + Regorafenib + AB928; Regorafenib (Control)
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of 21-day cycles, with the exception of the Atezolizumab + Selicrelumab + Bevacizumab, Atezolizumab + Idasanutlin, Atezolizumab + Regorafenib and Atezolizumab + Regorafenib + AB928 arms where the Atezolizumab will be administered by IV infusion every 2 weeks (Q2W) on Days 1 and 15 of each 28-day cycle.
  Arms: Atezolizumab + Idasanutlin; Atezolizumab + Imprime PGG + Bevacizumab; Atezolizumab + Isatuximab; Atezolizumab + LOAd703; Atezolizumab + Regorafenib; Atezolizumab + Regorafenib + AB928; Atezolizumab + Selicrelumab + Bevacizumab
Drug: Imprime PGG — Imprime PGG will be administered by IV infusion weekly on Days 1, 8, and 15 of each 21-day cycle.
  Arms: Atezolizumab + Imprime PGG + Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion on Day 1 of each 21-day cycle for the Atezolizumab + Imprime PGG + Bevacizumab arm, and on Day 1 and Day 15 of each 28-day cycle for the Atezolizumab + Selicrelumab + Bevacizumab arm.
  Arms: Atezolizumab + Imprime PGG + Bevacizumab; Atezolizumab + Selicrelumab + Bevacizumab
Drug: Isatuximab — Isatuximab will be administered on Day 1, 8 and 15 of cycle 1 and on day 1 of all subsequent cycles. Cycles will be 21 days long.
  Arms: Atezolizumab + Isatuximab
Drug: Selicrelumab — Selicrelumab will be administered by subcutaneous (SC) injection on Day 1 of cycles 1-4 and every third cycle thereafter. Cycles will be 28 days long.
  Arms: Atezolizumab + Selicrelumab + Bevacizumab
Drug: Idasanutlin — Idasanutlin will be administered orally on Days 1-5 of each 28-day cycle.
  Arms: Atezolizumab + Idasanutlin
Drug: AB928 — AB928 will be administered orally once daily on Days 1-28 of each 28-day cycle.
  Arms: Atezolizumab + Regorafenib + AB928
Genetic: LOAd703 — LOAd703 will be administered by intratumoral injection on Day 1 of each 21-day cycle.
  Other Names: Delolimogene mupadenorepvec
  Arms: Atezolizumab + LOAd703

SUMMARY:
A phase Ib/II, open-label, multicenter, randomized study designed to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of immunotherapy-based treatment combinations in patients with metastatic colorectal cancer (mCRC) that became refractory to first- and second-line standard therapies. Eligible patients will be assigned to one of several treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥ 3 months, as determined by the investigator
* Histologically confirmed adenocarcinoma originating from the colon or rectum
* Metastatic disease not amenable to local treatment
* Disease progression during or following not more than two separate lines of treatment for metastatic colorectal cancer (mCRC) that consisted of fluoropyrimidine-, oxaliplatin-, and irinotecan-containing chemotherapy in combination with a biologic agent
* Measurable disease (at least one target lesion) according to RECIST v1.1
* Adequate hematologic and end-organ function obtained within 14 days prior to initiation of study treatment

Exclusion Criteria:

* High microsatellite instability (MSI-H) tumor
* Presence of BRAFV600E mutation
* Prior treatment with any of the protocol-specified study treatments
* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Biologic treatment within 2 weeks prior to initiation of study treatment, or other systemic treatment for CRC within 2 weeks or 5 half-lives of the drug (whichever is shorter) prior to initiation of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Eligibility only for the control arm
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressant medication during study treatment
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the last dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Uncontrolled pleural effusion, pericardial effusion, ascites requiring recurrent drainage procedures (once monthly or more frequently), or tumor related-pain,
* Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected serum calcium >ULN)
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* History of malignancy other than CRC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Significant cardiovascular disease
* Grade ≥3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of severe allergic reactions to chimeric or humanized antibodies or fusion proteins
* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding
* Urine dipstick ≥ 2+ protein or ≥ 3.5 g of protein in a 24-hour urine collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Peter MacCallum Cancer Center, North Melbourne, Victoria, Australia
- France (4):
  - Centre Georges François Leclerc; Pharmacie des Essais Cliniques, Dijon
  - Centre Leon Berard, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy, Villejuif
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center., Seoul
- CHUV; Departement d'Oncologie, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 centers in 5 countries: United States, France, Republic of Korea, Australia, and Switzerland.
Period: Overall Study
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Started | 24 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Received at Least One Dose of Study Treatment (Safety Population) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 24 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Not completed — Death | 18 | 15 | 15 | 4 | 4 | 11 | 12 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized in the study, regardless of whether they actually received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703 | Total
Number analyzed (Participants) | 24 | 15 | 15 | 6 | 4 | 15 | 15 | 2 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (year) | 59.5 (10.3) | 57.8 (5.9) | 52.3 (12.0) | 66.8 (10.0) | 56.3 (6.8) | 56.4 (8.2) | 55.1 (9.2) | 58.0 (11.3) | 57.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 6 | 1 | 3 | 11 | 4 | 1 | 45
  Male | 12 | 8 | 9 | 5 | 1 | 4 | 11 | 1 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 3 | 1 | 0 | 1 | 0 | 1 | 12
  Not Hispanic or Latino | 21 | 10 | 11 | 4 | 4 | 11 | 14 | 1 | 76
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 7 | 6 | 4 | 0 | 1 | 5 | 8 | 0 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 15 | 7 | 10 | 5 | 3 | 7 | 6 | 2 | 55
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 6
ECOG score [Count of Participants; unit: Participants] — ECOG performance status scale. 0 - Fully active; able to carry on all predisease performance without restriction
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  Participants
    0 | 11 | 8 | 5 | 5 | 1 | 7 | 7 | 1 | 45
    1 | 13 | 7 | 10 | 1 | 3 | 8 | 8 | 1 | 51
Number of Metastatic Sites at Enrollment [Count of Participants; unit: Participants]
  1 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6
  2 | 4 | 5 | 3 | 3 | 3 | 7 | 5 | 0 | 30
  3 | 9 | 5 | 8 | 0 | 0 | 2 | 6 | 2 | 32
  >=4 | 8 | 4 | 4 | 3 | 1 | 5 | 3 | 0 | 28

OUTCOME MEASURES:

1. Primary Outcome: Best Confirmed Overall Response Rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: The best confirmed overall response rate (ORR) is defined as the percentage of participants with a complete response or partial response on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to RECIST v1.1. Participants could be classified as "Stable Disease" if the assessment was at least 6 weeks from randomization. Participants were classified as Missing if no post-baseline response assessments were available. Participants were classified as Not Evaluable if all post-baseline response assessments were unevaluable. The differences in ORR between the experimental arms and the corresponding control arm were calculated, along with 95% confidence intervals (CIs), using normal approximation of the binomial distribution. The 95% CIs for ORRs were constructed using the Clopper-Pearson method. The 95% CIs for the difference in rates were constructed using the Wald method with continuity correction.
Time Frame: From randomization until disease progression or loss of clinical benefit (up to 4 years)
Population: The efficacy evaluable population included all patients who received at least one dose of each drug for their assigned treatment regimen.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Percentage of Participants
  Responders (CR + PR) | 0 [0 to 17.65] | 0 [0 to 21.80] | 0 [0 to 21.80] | 0 [0 to 45.93] | 0 [0 to 60.24] | 6.7 [0.17 to 31.95] | 6.7 [0.17 to 31.95] | 0 [0 to 84.19]
  Complete Response (CR) | 0 [0 to 17.65] | 0 [0 to 21.80] | 0 [0 to 21.80] | 0 [0 to 45.93] | 0 [0 to 60.24] | 0 [0 to 21.80] | 0 [0 to 21.80] | 0 [0 to 84.19]
  Partial Response (PR) | 0 [0 to 17.65] | 0 [0 to 21.80] | 0 [0 to 21.80] | 0 [0 to 45.93] | 0 [0 to 60.24] | 6.7 [0.17 to 31.95] | 6.7 [0.17 to 31.95] | 0 [0 to 84.19]
  Stable Disease (SD) | 63.2 [38.36 to 83.71] | 33.3 [11.82 to 61.62] | 20.0 [4.33 to 48.09] | 50 [11.81 to 88.19] | 0 [0 to 60.24] | 33.3 [11.82 to 61.62] | 53.3 [26.59 to 78.73] | 0 [0 to 84.19]
  Progressive Disease (PD) | 26.3 [9.15 to 51.20] | 66.7 [38.38 to 88.18] | 66.7 [38.38 to 88.18] | 33.3 [4.33 to 77.72] | 100 [39.76 to 100] | 46.7 [21.27 to 73.41] | 26.7 [7.79 to 55.10] | 100 [15.81 to 100]
  Not Evaluable | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 13.3 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 13.3 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing.
  Missing | 10.5 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 16.7 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 13.3 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing. | 0 [NA to NA] — The 95% CI was only calculated for responses per RECIST, not for participants who were not evaluable or missing.
Statistical Analysis 1: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Test type: Other; Difference in Overall Response Rate = 6.67, 95% CI 2-sided [-11.92 to 25.25] — The difference in ORR was calculated as the experimental arm (Atezolizumab + Regorafenib) subtracted from the control arm (Regorafenib)
Statistical Analysis 2: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Test type: Other; Difference in Overall Response Rate = 6.67, 95% CI 2-sided [-11.92 to 25.25] — The difference in ORR was calculated as the experimental arm (Atezolizumab + Regorafenib + AB928) subtracted from the control arm (Regorafenib)

2. Secondary Outcome: Progression-Free Survival (PFS) as Determined by Investigator According to RECIST v1.1
Description: Progression-free survival (PFS) after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), was determined by the investigator according to RECIST v1.1. For participants who did not have documented disease progression or death, PFS was censored at the day of the last tumor assessment. The Kaplan-Meier method was used to estimate the median for PFS with 95% confidence intervals (CIs) constructed through use of the Brookmeyer and Crowley method.
Time Frame: From randomization up to the first occurrence of disease or death from any cause (up to 4 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Months | 2.83 [2.20 to 3.02] | 1.51 [1.38 to 2.79] | 1.41 [1.41 to 1.77] | 4.21 [1.68 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred. | 1.26 [0.82 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred. | 1.81 [1.38 to 2.96] | 4.60 [2.60 to 5.78] | 1.58 [1.51 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred.
Statistical Analysis 1: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Test type: Other; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.67 to 2.73]
Statistical Analysis 2: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Test type: Other; Hazard Ratio (HR) = 2.30, 95% CI 2-sided [1.08 to 4.88]
Statistical Analysis 3: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Test type: Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.29 to 2.18]
Statistical Analysis 4: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Test type: Other; Hazard Ratio (HR) = 2.00, 95% CI 2-sided [0.64 to 6.24]
Statistical Analysis 5: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Test type: Other; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [0.83 to 3.63]
Statistical Analysis 6: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Test type: Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.39 to 1.63]
Statistical Analysis 7: Comparison: Regorafenib (Control) vs Atezolizumab + LOAd703; Test type: Other; Hazard Ratio (HR) = 5.64, 95% CI 2-sided [0.94 to 33.82]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. The Kaplan-Meier method was used to estimate the median for OS with 95% confidence intervals (CIs) constructed through use of the Brookmeyer and Crowley method.
Time Frame: From randomization up to death from any cause (up to 4 years)
Population: The efficacy evaluable population included all participants who received at least one dose of each study drug for their assigned treatment regimen.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Months | 10.15 [4.40 to 12.29] | 5.72 [4.37 to 10.51] | 5.13 [3.12 to 7.75] | 14.36 [3.22 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred. | 5.93 [1.61 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred. | 11.01 [5.29 to 16.66] | 8.67 [6.60 to 14.62] | 4.07 [NA to NA] — The lower and upper limits of the 95% CI were not estimable because too few events had occurred.
Statistical Analysis 1: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Atezolizumab + Imprime PGG + Bevacizumab vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.71 to 2.93]
Statistical Analysis 2: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Atezolizumab + Isatuximab vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.68 to 2.81]
Statistical Analysis 3: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Atezolizumab + Selicrelumab + Bevacizumab vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.30 to 2.72]
Statistical Analysis 4: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Atezolizumab + Idasanutlin vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.42 to 3.84]
Statistical Analysis 5: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Atezolizumab + Regorafenib vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.39 to 1.88]
Statistical Analysis 6: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Atezolizumab + Regorafenib + AB928 vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.43 to 1.96]
Statistical Analysis 7: Comparison: Regorafenib (Control) vs Atezolizumab + LOAd703; Atezolizumab + LOAd703 vs. Regorafenib (Control) Hazard Ratio for OS; Test type: Other — Kaplan-Meier; Hazard Ratio (HR) = 2.88, 95% CI 2-sided [0.33 to 24.85]

4. Secondary Outcome: Percentage of Participants Who Were Alive at Landmark Timepoints for Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. OS is shown as the percentage of participants who were event-free at the landmark timepoints of 3, 6, 12, and 18 months.
Time Frame: 3, 6, 12, and 18 months
Population: The efficacy evaluable population included all participants who received at least one dose of each study drug for their assigned treatment regimen. The number analyzed at each landmark timepoint indicates the number of participants who were remaining at risk for an event. The event-free rate was not estimable (NE) for landmark timepoints at which 0 participants were remaining at risk for an an event.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Percentage of Participants
  3 Months: number analyzed (Participants) | 16 | 15 | 11 | 5 | 3 | 11 | 13 | 1
  3 Months | 84.21 [67.81 to 100] | 100.00 [100.00 to 100.00] | 73.33 [50.95 to 95.71] | 100.00 [100.00 to 100.00] | 75.00 [32.57 to 100.00] | 78.97 [57.78 to 100.00] | 86.67 [69.46 to 100.00] | 100.00 [100.00 to 100.00]
  6 Months: number analyzed (Participants) | 11 | 7 | 6 | 3 | 2 | 10 | 11 | 0
  6 Months | 63.16 [41.47 to 84.85] | 46.67 [21.42 to 71.91] | 40.00 [15.21 to 64.79] | 80.00 [44.94 to 100.00] | 50.00 [1.00 to 99.00] | 71.79 [48.32 to 95.27] | 73.33 [50.95 to 95.71] |
  12 Months: number analyzed (Participants) | 6 | 3 | 4 | 2 | 1 | 5 | 5 | 0
  12 Months | 34.45 [12.42 to 56.48] | 20.00 [0.00 to 40.24] | 26.67 [4.29 to 49.05] | 53.33 [4.68 to 100] | 25.00 [0.00 to 67.43] | 39.89 [13.18 to 66.59] | 33.33 [9.48 to 57.19] |
  18 Months: number analyzed (Participants) | 3 | 1 | 3 | 1 | 1 | 3 | 4 | 0
  18 Months | 17.22 [0.00 to 34.87] | 6.67 [0.00 to 19.29] | 20.00 [0.00 to 40.24] | 26.67 [0.00 to 70.97] | 25.00 [0.00 to 67.43] | 23.93 [0.48 to 47.39] | 26.67 [4.29 to 49.05] |
Statistical Analysis 1: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Difference in OS event-free rate at 3 months for the Atezolizumab + Imprime PGG + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 15.79, 95% CI 2-sided [-0.61 to 32.19]
Statistical Analysis 2: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Difference in OS event-free rate at 6 months for the Atezolizumab + Imprime PGG + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -16.49, 95% CI 2-sided [-49.78 to 16.79]
Statistical Analysis 3: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Difference in OS event-free rate at 12 months for the Atezolizumab + Imprime PGG + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -14.45, 95% CI 2-sided [-44.37 to 15.47]
Statistical Analysis 4: Comparison: Regorafenib (Control) vs Atezolizumab + Imprime PGG + Bevacizumab; Difference in OS event-free rate at 18 months for the Atezolizumab + Imprime PGG + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -10.56, 95% CI 2-sided [-32.25 to 11.14]
Statistical Analysis 5: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Difference in OS event-free rate at 3 months for the Atezolizumab + Isatuximab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -10.88, 95% CI 2-sided [-38.62 to 16.87]
Statistical Analysis 6: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Difference in OS event-free rate at 6 months for the Atezolizumab + Isatuximab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -23.16, 95% CI 2-sided [-56.10 to 9.78]
Statistical Analysis 7: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Difference in OS event-free rate at 12 months for the Atezolizumab + Isatuximab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -7.78, 95% CI 2-sided [-39.19 to 23.62]
Statistical Analysis 8: Comparison: Regorafenib (Control) vs Atezolizumab + Isatuximab; Difference in OS event-free rate at 18 months for the Atezolizumab + Isatuximab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 2.78, 95% CI 2-sided [-24.08 to 29.63]
Statistical Analysis 9: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Difference in OS event-free rate at 3 months for the Atezolizumab + Selicrelumab + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 15.79, 95% CI 2-sided [-0.61 to 32.19]
Statistical Analysis 10: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Difference in OS event-free rate at 6 months for the Atezolizumab + Selicrelumab + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 16.84, 95% CI 2-sided [-24.39 to 58.07]
Statistical Analysis 11: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Difference in OS event-free rate at 12 months for the Atezolizumab + Selicrelumab + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 18.88, 95% CI 2-sided [-34.53 to 72.30]
Statistical Analysis 12: Comparison: Regorafenib (Control) vs Atezolizumab + Selicrelumab + Bevacizumab; Difference in OS event-free rate at 18 months for the Atezolizumab + Selicrelumab + Bevacizumab vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 9.44, 95% CI 2-sided [-38.19 to 57.08]
Statistical Analysis 13: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Difference in OS event-free rate at 3 months for the Atezolizumab + Idasanutlin vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -9.21, 95% CI 2-sided [-54.70 to 36.28]
Statistical Analysis 14: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Difference in OS event-free rate at 6 months for the Atezolizumab + Idasanutlin vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -13.16, 95% CI 2-sided [-66.74 to 40.43]
Statistical Analysis 15: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Difference in OS event-free rate at 12 months for the Atezolizumab + Idasanutlin vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -9.45, 95% CI 2-sided [-57.26 to 38.36]
Statistical Analysis 16: Comparison: Regorafenib (Control) vs Atezolizumab + Idasanutlin; Difference in OS event-free rate at 18 months for the Atezolizumab + Idasanutlin vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 7.78, 95% CI 2-sided [-38.18 to 53.73]
Statistical Analysis 17: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Difference in OS event-free rate at 3 months for the Atezolizumab + Regorafenib vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -5.24, 95% CI 2-sided [-32.03 to 21.56]
Statistical Analysis 18: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Difference in OS event-free rate at 6 months for the Atezolizumab + Regorafenib vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 8.64, 95% CI 2-sided [-23.33 to 40.60]
Statistical Analysis 19: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Difference in OS event-free rate at 12 months for the Atezolizumab + Regorafenib vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 5.44, 95% CI 2-sided [-29.19 to 40.06]
Statistical Analysis 20: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib; Difference in OS event-free rate at 18 months for the Atezolizumab + Regorafenib vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 6.71, 95% CI 2-sided [-22.64 to 36.06]
Statistical Analysis 21: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Difference in OS event-free rate at 3 months for the Atezolizumab + Regorafenib + AB928 vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 2.46, 95% CI 2-sided [-21.31 to 26.22]
Statistical Analysis 22: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Difference in OS event-free rate at 6 months for the Atezolizumab + Regorafenib + AB928 vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 10.18, 95% CI 2-sided [-20.99 to 41.34]
Statistical Analysis 23: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Difference in OS event-free rate at 12 months for the Atezolizumab + Regorafenib + AB928 vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = -1.12, 95% CI 2-sided [-33.59 to 31.36]
Statistical Analysis 24: Comparison: Regorafenib (Control) vs Atezolizumab + Regorafenib + AB928; Difference in OS event-free rate at 18 months for the Atezolizumab + Regorafenib + AB928 vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 9.44, 95% CI 2-sided [-19.06 to 37.94]
Statistical Analysis 25: Comparison: Regorafenib (Control) vs Atezolizumab + LOAd703; Difference in OS event-free rate at 3 months for the Atezolizumab +LOAd703 vs. Regorafenib (Control) arms; Test type: Other; Difference in OS Event-Free Rate = 15.79, 95% CI 2-sided [-0.61 to 32.19]

5. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1
Description: Duration of response is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause.
Time Frame: From the date of first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 4 years)
Population: The duration of response analysis included all participants from the efficacy evaluable population who had a confirmed overall response; only 1 participant in each of the atezolizumab + regorafenib arm and the atezolizumab + regorafenib + AB928 arm had a confirmed response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Months |  |  |  |  |  | 3.12 [NA to NA] — Only 1 participant had a confirmed response; 95% CI could not be calculated. | 5.75 [NA to NA] — Only 1 participant had a confirmed response; 95% CI could not be calculated. |

6. Secondary Outcome: Disease Control Rate (DCR), as Determined by the Investigator Per RECIST v1.1
Description: Disease control rate is defined as the percentage of participants with stable disease for ≥12 weeks or a complete or partial response, as determined by the investigator according to RECIST v1.1.
Time Frame: From randomization until disease progression or loss of clinical benefit (up to 4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Percentage of Participants | 15.8 [3.38 to 39.58] | 13.3 [1.66 to 40.46] | 6.7 [0.17 to 31.95] | 33.3 [4.33 to 77.72] | 0 [0.00 to 60.24] | 13.3 [1.66 to 40.46] | 40.0 [16.34 to 67.71] | 0 [0.00 to 84.19]

7. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: The incidence, nature, and severity of adverse events (AEs) are reported, with severity determined according to NCI CTCAE v4.0. All AEs were reported until 30 days after the last study dose or until start of new systemic anti-cancer therapy. Serious AEs and AEs of special interest were reported until 135 days (or 180 days for the Atezolizumab + LOAd703 arm only) after the last dose of study treatment.
Time Frame: Adverse event data were collected from baseline up to 6 months after the last dose of study treatment (up to 640 days); deaths (all-cause) were reported from baseline through survival follow-up (up to 4 years)
Population: The safety-evaluable population included all patients who received any amount of dose of any component of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
Number analyzed (Participants) | 19 | 15 | 15 | 6 | 4 | 15 | 15 | 2
Percentage of Participants
  Adverse Event (AE) | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100
  Death | 89.5 | 100 | 100 | 66.7 | 100 | 73.3 | 80.0 | 50.0
  Withdrawn from Stage due to an AE | 15.8 | 6.7 | 0 | 0 | 0 | 6.7 | 6.7 | 0
  AE with a Fatal Outcome | 10.5 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0
  Serious AE (SAE) | 26.3 | 6.7 | 33.3 | 50.0 | 25.0 | 46.7 | 46.7 | 50.0
  SAE Leading to Withdrawal from any Treatment | 21.1 | 6.7 | 0 | 0 | 0 | 6.7 | 0 | 0
  SAE Leading to Dose Modification/Interruption | 5.3 | 0 | 6.7 | 50.0 | 0 | 26.7 | 46.7 | 0
  Related SAE | 5.3 | 6.7 | 0 | 50.0 | 25.0 | 26.7 | 33.3 | 50.0
  AE Leading to Withdrawal from any Treatment | 26.3 | 6.7 | 0 | 0 | 0 | 20.0 | 6.7 | 0
  AE Leading to Dose Modification/Interruption | 63.2 | 40.0 | 13.3 | 50.0 | 75.0 | 86.7 | 93.3 | 0
  Related AE | 94.7 | 86.7 | 86.7 | 100 | 100 | 93.3 | 100 | 50.0
  Related AE Leading to Withdrawal from any Treatment | 10.5 | 6.7 | 0 | 0 | 0 | 6.7 | 6.7 | 0
  Related AE Leading to Dose Modification/Interruption | 47.4 | 33.3 | 0 | 33.3 | 75.0 | 73.3 | 93.3 | 0
  Grade 3-5 AE | 68.4 | 20.0 | 46.7 | 50.0 | 75.0 | 66.7 | 60.0 | 0
  Worst Grade AE: 5 | 10.5 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0
  Worst Grade AE: 4 | 5.3 | 0 | 6.7 | 0 | 25.0 | 6.7 | 13.3 | 0
  Worst Grade AE: 3 | 52.6 | 20.0 | 40.0 | 50.0 | 50.0 | 53.3 | 46.7 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from first study dose up to 6 months after the last dose of study treatment (up to 640 days); deaths (all-cause) were reported from enrolment through survival follow-up (up to 4 years).
Description: All-Cause Mortality is reported in the all-enrolled patients population. Adverse events (AEs) are reported in the safety population, defined as all those who received ≥1 dose of study treatment. One participant in the Regorafenib arm died before receiving study dose. All AEs were reported until 30 days after the last study dose or until the start of new systemic anti-cancer therapy. Serious AEs and AEs of special interest are reported until up to 180 days after last study dose.
Arm/Group | Regorafenib (Control) | Atezolizumab + Imprime PGG + Bevacizumab | Atezolizumab + Isatuximab | Atezolizumab + Selicrelumab + Bevacizumab | Atezolizumab + Idasanutlin | Atezolizumab + Regorafenib | Atezolizumab + Regorafenib + AB928 | Atezolizumab + LOAd703
All-Cause Mortality (participants affected / at risk) | 18/24 | 15/15 | 15/15 | 4/6 | 4/4 | 11/15 | 12/15 | 1/2
Serious Adverse Events (participants affected / at risk) | 5/19 | 1/15 | 5/15 | 3/6 | 1/4 | 7/15 | 7/15 | 1/2
Other Adverse Events (participants affected / at risk) | 19/19 | 15/15 | 15/15 | 6/6 | 4/4 | 15/15 | 15/15 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Control) (N=19) | Atezolizumab + Imprime PGG + Bevacizumab (N=15) | Atezolizumab + Isatuximab (N=15) | Atezolizumab + Selicrelumab + Bevacizumab (N=6) | Atezolizumab + Idasanutlin (N=4) | Atezolizumab + Regorafenib (N=15) | Atezolizumab + Regorafenib + AB928 (N=15) | Atezolizumab + LOAd703 (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perforation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Control) (N=19) | Atezolizumab + Imprime PGG + Bevacizumab (N=15) | Atezolizumab + Isatuximab (N=15) | Atezolizumab + Selicrelumab + Bevacizumab (N=6) | Atezolizumab + Idasanutlin (N=4) | Atezolizumab + Regorafenib (N=15) | Atezolizumab + Regorafenib + AB928 (N=15) | Atezolizumab + LOAd703 (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 1 (2) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 6 (9) | 2 (3) | 2 (2) | 2 (4) | 7 (8) | 4 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (5) | 6 (8) | 0 (0) | 4 (11) | 3 (3) | 2 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (7) | 3 (4) | 1 (1) | 4 (6) | 3 (4) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 4 (4) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (8) | 7 (11) | 9 (11) | 2 (2) | 1 (2) | 7 (8) | 4 (6) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 7 (9) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 8 (16) | 11 (13) | 0 (0) | 0 (0) | 2 (2) | 4 (7) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site rash (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 5 (6) | 4 (4) | 2 (2) | 1 (1) | 6 (6) | 5 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 4 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 6 (8) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (7) | 3 (3) | 1 (1) | 1 (5) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study is not designed to make explicit power and Type I error considerations for a hypothesis test. Instead, this study is designed to obtain preliminary efficacy, safety, and PK data. No formal statistical hypothesis testing was performed in this study. Due to the limited sample size, the results need to be interpreted with caution. For the Atezo+Idasa and Atezo+LOAd703 groups, no meaningful conclusion could be drawn because these experimental arms have been terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03555149/Prot_SAP_000.pdf